CLINICAL TRIAL: NCT05894434
Title: Ameliorating Stroke-induced Hemianopia Via Multisensory Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00093457
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-03

CONDITIONS: Hemianopia, Homonymous; Cortical Blindness, Unspecified Side of Brain
Keywords: multisensory; visual perception; neurorehabilitation
MeSH Terms: conditions — Hemianopsia; Blindness, Cortical

STUDY DESIGN:
Intervention Model Description: There are two principal sub-studies: standard intervention and early intervention. Each sub-study contains a multisensory training group (experimental arm) and a unisensory training group (control arm). The unisensory training group crosses over to multisensory training at its completion. Thus, the model design is both factorial and crossover.
Who Masked: Outcomes Assessor
Masking Description: The experimental and control paradigms are based on sensory stimulation and there is no practical way to mask the participant from its nature, although they are not informed as to what the expected results will be. The outcomes assessor will be blinded to which stimulation arm preceded the data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Intervention: Multisensory Training (Experimental): Patients with stable hemianopia (>6 months) are given multisensory training
  Interventions: Behavioral: Multisensory Training
- Standard Intervention: Unisensory Training (Active Comparator): Patients with stable hemianopia (>6 months) are given auditory training and crossover to multisensory training
  Interventions: Behavioral: Multisensory Training; Behavioral: Unisensory Training
- Early Intervention: Multisensory Training (Experimental): Patients with early hemianopia (<1 months) are given multisensory training
  Interventions: Behavioral: Multisensory Training
- Early Intervention: Unisensory Training (Active Comparator): Patients with early hemianopia (<1 months) are given auditory training and crossover to multisensory training
  Interventions: Behavioral: Multisensory Training; Behavioral: Unisensory Training

INTERVENTIONS:
Behavioral: Multisensory Training — The procedure involves repeatedly presenting identical visual-auditory stimuli at a single location in the hemianopic field (initially at 45° of eccentricity along the azimuth) while the patient maintains central fixation (0°, 0°). The visual (a 500 ms flash) and auditory (500 ms broadband noise burst) stimuli are in spatial and temporal congruence.
Behavioral: Unisensory Training — The procedure involves repeatedly presenting identical auditory stimuli (500 ms broadband noise burst) at a single location in the hemianopic field (initially at 45° of eccentricity along the azimuth) while the patient maintains central fixation (0°, 0°).
  Arms: Early Intervention: Unisensory Training; Standard Intervention: Unisensory Training

SUMMARY:
This study seeks to determine the extent of the visual capabilities that can be restored in hemianopic stroke patients by a multisensory training technique and evaluate changes in the brain that the training induces. The effectiveness of the technique will be evaluated in two interventional contexts: patients whose blindness is long-standing and stable, and another in which intervention is as soon as possible after the stroke.

DETAILED DESCRIPTION:
The aims of the study are to:

1. To identify the visual capabilities and neural circuits in stroke patients with stable hemianopia (>6 months) that recover after regular multisensory (vs. unisensory) training sessions. This involves:

1A. Using clinical ophthalmological tests and visual perceptual tests to evaluate the visual capabilities that are recovered.

1B. Determining whether the size or extent of cortical lesions are predictive of changes induced by the training technique, and tracking changes in the residual visual circuits using functional magnetic resonance imaging (fMRI).

1C. Determining if the training-induced changes improve, persist, or degrade over time by re-assessment at a 12-month followup.

2. Evaluate the effectiveness of an earlier (<1 month post-stroke) and more intense training intervention strategy using the above approach and comparing the outcomes in these two approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Homonymous hemianopia diagnosed and referred by a neurologist, confirmed with Humphrey test (Goldmann size V) on first visit. Hemianopia must have been evident for at least 6 months for inclusion in the first experiment and <1 month for inclusion in the second
* Cognitively normal, defined as having normal activities of daily living OR has received a cognitive adjudication of normal through the Wake Forest University School of Medicine or equivalent within the past 12 months
* MRI compatible
* Has reliable transportation or is able to use transportation provided by the study
* English speaking

Exclusion Criteria:

* Current major medical problems that might independently affect cognition, vision, or interfere with ability to attend study visits. This includes pathology of the retina or optic nerve explanatory of blindness
* Unable or unwilling to attend scheduled testing and training sessions, including the 12 month follow up
* Current diagnosis of a major neurological disorder that could interfere with the ability to follow task instructions (Dementia, Parkinson's disease, etc.) or that may interfere with the rehabilitation paradigm (uncorrected asymmetric hearing loss, deafness, hemineglect)
* Unwilling or unable to provide consent for study participation
* Current stroke symptoms deemed exclusionary by a study physician. This will be reviewed on a case-by-case basis by a study physician to determine whether factors may affect study outcomes, aims, or integrity
* Taking medication that could negatively influence safety during the intervention
* Enrolled in another interventional research study <= 3 months prior to beginning this study
* Self-reports regularly drinking > 14 alcoholic beverages a week or current illicit drug use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Clinical Ophthalmological Test Scores | Baseline
  Humphrey tests - The Humphrey visual field test measures the entire area of peripheral vision that can be seen while the eye is focused on a central point. During this test, lights of varying intensities appear in different parts of the visual field while the patient's eye is focused on a certain spot. A normal visual field extends approximately 100° temporally (laterally), 60° nasally, 60° superiorly, and 70° inferiorly. A normal visual field measures about: 90 degrees temporally. 50 degrees superiorly and nasally. 60 degrees inferiorly
Clinical Ophthalmological Test Scores | Day 15
  Humphrey tests - The Humphrey visual field test measures the entire area of peripheral vision that can be seen while the eye is focused on a central point. During this test, lights of varying intensities appear in different parts of the visual field while the patient's eye is focused on a certain spot. A normal visual field extends approximately 100° temporally (laterally), 60° nasally, 60° superiorly, and 70° inferiorly. A normal visual field measures about: 90 degrees temporally. 50 degrees superiorly and nasally. 60 degrees inferiorly
Clinical Ophthalmological Test Scores | Week 8
  Humphrey tests - The Humphrey visual field test measures the entire area of peripheral vision that can be seen while the eye is focused on a central point. During this test, lights of varying intensities appear in different parts of the visual field while the patient's eye is focused on a certain spot. A normal visual field extends approximately 100° temporally (laterally), 60° nasally, 60° superiorly, and 70° inferiorly. A normal visual field measures about: 90 degrees temporally. 50 degrees superiorly and nasally. 60 degrees inferiorly
Clinical Ophthalmological Test Scores | Week 10
  Humphrey tests - The Humphrey visual field test measures the entire area of peripheral vision that can be seen while the eye is focused on a central point. During this test, lights of varying intensities appear in different parts of the visual field while the patient's eye is focused on a certain spot. A normal visual field extends approximately 100° temporally (laterally), 60° nasally, 60° superiorly, and 70° inferiorly. A normal visual field measures about: 90 degrees temporally. 50 degrees superiorly and nasally. 60 degrees inferiorly
Clinical Ophthalmological Test Scores | Week 16
  Humphrey tests - The Humphrey visual field test measures the entire area of peripheral vision that can be seen while the eye is focused on a central point. During this test, lights of varying intensities appear in different parts of the visual field while the patient's eye is focused on a certain spot. A normal visual field extends approximately 100° temporally (laterally), 60° nasally, 60° superiorly, and 70° inferiorly. A normal visual field measures about: 90 degrees temporally. 50 degrees superiorly and nasally. 60 degrees inferiorly
Clinical Ophthalmological Test Scores | Week 48
  Humphrey tests - The Humphrey visual field test measures the entire area of peripheral vision that can be seen while the eye is focused on a central point. During this test, lights of varying intensities appear in different parts of the visual field while the patient's eye is focused on a certain spot. A normal visual field extends approximately 100° temporally (laterally), 60° nasally, 60° superiorly, and 70° inferiorly. A normal visual field measures about: 90 degrees temporally. 50 degrees superiorly and nasally. 60 degrees inferiorly
Clinical Ophthalmological Test Scores | Week 50
  Humphrey tests - The Humphrey visual field test measures the entire area of peripheral vision that can be seen while the eye is focused on a central point. During this test, lights of varying intensities appear in different parts of the visual field while the patient's eye is focused on a certain spot. A normal visual field extends approximately 100° temporally (laterally), 60° nasally, 60° superiorly, and 70° inferiorly. A normal visual field measures about: 90 degrees temporally. 50 degrees superiorly and nasally. 60 degrees inferiorly
Clinical Ophthalmological Test Scores | Week 56
  Humphrey tests - The Humphrey visual field test measures the entire area of peripheral vision that can be seen while the eye is focused on a central point. During this test, lights of varying intensities appear in different parts of the visual field while the patient's eye is focused on a certain spot. A normal visual field extends approximately 100° temporally (laterally), 60° nasally, 60° superiorly, and 70° inferiorly. A normal visual field measures about: 90 degrees temporally. 50 degrees superiorly and nasally. 60 degrees inferiorly
Clinical Ophthalmological Test Scores | Week 64
  Humphrey tests - The Humphrey visual field test measures the entire area of peripheral vision that can be seen while the eye is focused on a central point. During this test, lights of varying intensities appear in different parts of the visual field while the patient's eye is focused on a certain spot. A normal visual field extends approximately 100° temporally (laterally), 60° nasally, 60° superiorly, and 70° inferiorly. A normal visual field measures about: 90 degrees temporally. 50 degrees superiorly and nasally. 60 degrees inferiorly
Visual Perception Test Scores | Baseline
  Ability to detect and discriminate different visual features - The participant is asked to indicate (via button press) whether the test stimulus matches the sample (left button), does not match the sample (right button), or there was no test stimulus (withhold response).
Visual Perception Test Scores | Day 15
  Ability to detect and discriminate different visual features - The participant is asked to indicate (via button press) whether the test stimulus matches the sample (left button), does not match the sample (right button), or there was no test stimulus (withhold response).
Visual Perception Test Scores | Week 8
  Ability to detect and discriminate different visual features - The participant is asked to indicate (via button press) whether the test stimulus matches the sample (left button), does not match the sample (right button), or there was no test stimulus (withhold response).
Visual Perception Test Scores | Week 10
  Ability to detect and discriminate different visual features - The participant is asked to indicate (via button press) whether the test stimulus matches the sample (left button), does not match the sample (right button), or there was no test stimulus (withhold response).
Visual Perception Test Scores | Week 16
  Ability to detect and discriminate different visual features - The participant is asked to indicate (via button press) whether the test stimulus matches the sample (left button), does not match the sample (right button), or there was no test stimulus (withhold response).
Visual Perception Test Scores | Week 48
  Ability to detect and discriminate different visual features - The participant is asked to indicate (via button press) whether the test stimulus matches the sample (left button), does not match the sample (right button), or there was no test stimulus (withhold response).
Visual Perception Test Scores | Week 50
  Ability to detect and discriminate different visual features - The participant is asked to indicate (via button press) whether the test stimulus matches the sample (left button), does not match the sample (right button), or there was no test stimulus (withhold response).
Visual Perception Test Scores | Week 56
  Ability to detect and discriminate different visual features - The participant is asked to indicate (via button press) whether the test stimulus matches the sample (left button), does not match the sample (right button), or there was no test stimulus (withhold response).
Visual Perception Test Scores | Week 64
  Ability to detect and discriminate different visual features - The participant is asked to indicate (via button press) whether the test stimulus matches the sample (left button), does not match the sample (right button), or there was no test stimulus (withhold response).
Functional magnetic resonance imaging (fMRI) scans | Baseline
  Used to measure functional lesion and assess changes - fMRI enables the detection of abnormalities of the brain, as well as the assessment of the normal functional anatomy of the brain, which cannot be accomplished with other imaging techniques.
Functional magnetic resonance imaging (fMRI) scans | Day 15
  Used to measure functional lesion and assess changes - fMRI enables the detection of abnormalities of the brain, as well as the assessment of the normal functional anatomy of the brain, which cannot be accomplished with other imaging techniques.
Functional magnetic resonance imaging (fMRI) scans | Week 8
  Used to measure functional lesion and assess changes - fMRI enables the detection of abnormalities of the brain, as well as the assessment of the normal functional anatomy of the brain, which cannot be accomplished with other imaging techniques.
Functional magnetic resonance imaging (fMRI) scans | Week 10
  Used to measure functional lesion and assess changes - fMRI enables the detection of abnormalities of the brain, as well as the assessment of the normal functional anatomy of the brain, which cannot be accomplished with other imaging techniques.
Functional magnetic resonance imaging (fMRI) scans | Week 16
  Used to measure functional lesion and assess changes - fMRI enables the detection of abnormalities of the brain, as well as the assessment of the normal functional anatomy of the brain, which cannot be accomplished with other imaging techniques.
Functional magnetic resonance imaging (fMRI) scans | Week 48
  Used to measure functional lesion and assess changes - fMRI enables the detection of abnormalities of the brain, as well as the assessment of the normal functional anatomy of the brain, which cannot be accomplished with other imaging techniques.
Functional magnetic resonance imaging (fMRI) scans | Week 50
  Used to measure functional lesion and assess changes - fMRI enables the detection of abnormalities of the brain, as well as the assessment of the normal functional anatomy of the brain, which cannot be accomplished with other imaging techniques.
Functional magnetic resonance imaging (fMRI) scans | Week 56
  Used to measure functional lesion and assess changes - fMRI enables the detection of abnormalities of the brain, as well as the assessment of the normal functional anatomy of the brain, which cannot be accomplished with other imaging techniques.
Functional magnetic resonance imaging (fMRI) scans | Week 64
  Used to measure functional lesion and assess changes - fMRI enables the detection of abnormalities of the brain, as well as the assessment of the normal functional anatomy of the brain, which cannot be accomplished with other imaging techniques.
Quality of Life (QoL) Assessment | Baseline
  The Veterans Affairs Low-Vision Visual Functioning Questionnaire-48 (VA-LV-VFQ-48) - A higher score on the VA LV VFQ-48 indicates better ability or less difficulty in performing activities
Quality of Life (QoL) Assessment | Day 15
  The Veterans Affairs Low-Vision Visual Functioning Questionnaire-48 (VA-LV-VFQ-48) - A higher score on the VA LV VFQ-48 indicates better ability or less difficulty in performing activities
Quality of Life (QoL) Assessment | Week 8
  The Veterans Affairs Low-Vision Visual Functioning Questionnaire-48 (VA-LV-VFQ-48) - A higher score on the VA LV VFQ-48 indicates better ability or less difficulty in performing activities
Quality of Life (QoL) Assessment | Week 10
  The Veterans Affairs Low-Vision Visual Functioning Questionnaire-48 (VA-LV-VFQ-48) - A higher score on the VA LV VFQ-48 indicates better ability or less difficulty in performing activities
Quality of Life (QoL) Assessment | Week 16
  The Veterans Affairs Low-Vision Visual Functioning Questionnaire-48 (VA-LV-VFQ-48) - A higher score on the VA LV VFQ-48 indicates better ability or less difficulty in performing activities
Quality of Life (QoL) Assessment | Week 48
  The Veterans Affairs Low-Vision Visual Functioning Questionnaire-48 (VA-LV-VFQ-48) - A higher score on the VA LV VFQ-48 indicates better ability or less difficulty in performing activities
Quality of Life (QoL) Assessment | Week 50
  The Veterans Affairs Low-Vision Visual Functioning Questionnaire-48 (VA-LV-VFQ-48) - A higher score on the VA LV VFQ-48 indicates better ability or less difficulty in performing activities
Quality of Life (QoL) Assessment | Week 56
  The Veterans Affairs Low-Vision Visual Functioning Questionnaire-48 (VA-LV-VFQ-48) - A higher score on the VA LV VFQ-48 indicates better ability or less difficulty in performing activities
Quality of Life (QoL) Assessment | Week 64
  The Veterans Affairs Low-Vision Visual Functioning Questionnaire-48 (VA-LV-VFQ-48) - A higher score on the VA LV VFQ-48 indicates better ability or less difficulty in performing activities

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin A Rowland, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Published data from the project will be made available to other researchers via the NIMH NDA repository. This may or may not include IPD.